CLINICAL TRIAL: NCT00317967
Title: Statin Induced Regression of Cardiomyopathy Trial - SirCat
Brief Title: Study to Determine if Atorvastatin Reduces Size and Stiffness of Muscle in the Left Ventricle of the Heart
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Dr. Bob Sheldon, Professor of Cardiac Sciences, Medicine and Medical Genetics, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-Sheldon
Record Dates: First submitted 2006-04-24; First posted 2006-04-25 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Hypertrophic cardiomyopathy; Statin therapy; Regression; Heart failure; Arrhythmias; Sudden cardiac death
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Heart Failure; Arrhythmias, Cardiac; Death, Sudden, Cardiac | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Atorvastatin
  Interventions: Drug: Atorvastatin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 80 mg pills daily
  Arms: 1
Drug: Placebo — 80 mg pills daily
  Arms: 2

SUMMARY:
The purpose of this study is to determine if a drug called atorvastatin will reduce the size and stiffness of the muscle in the left ventricle of the heart.

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is a primary disorder of the heart characterized by a thickened, fibrotic myocardium, with or without a dynamic left ventricular outflow tract gradient. It is a common heritable cardiovascular disease, with a population prevalence of 0.1% to 0.2%. Symptoms of congestive heart failure are extremely common in patients with HCM. Progression to disabling and debilitating symptoms [New York Heart Association (NYHA) class III and IV] is relatively common, occurring in 15% to 20% of unselected populations. The rate of progression to NYHA class III or IV or death from heart failure or stroke is high, with a relative risk 2.7. Management of symptoms can be very challenging, involve multiple medications, and 5% of patients may develop drug refractory heart failure, requiring invasive intervention. HCM is the most common cause of sudden death among young competitive athletes. Ventricular tachyarrhythmias appear to be the primary mechanism; however, other arrhythmias involved include asystole, rapid atrial fibrillation, and electrical mechanical dissociation. Patients may develop progressive myocardial wall thinning, a reduction in systolic performance, and an increase in left ventricular dimensions. Progressive wall thinning may be especially common in patients with initially severe hypertrophy. There is no cure for this condition. There is now evidence from both animal and human studies of a treatment that promises to reverse hypertrophy - HMG CoA reductase inhibitors. Clearly, studies of treatments that might cause regression of hypertrophy are timely and important.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over with HCM in the absence of another cardiac or systemic disease capable of producing a prespecified wall thickening

Exclusion Criteria:

* Required use of statin therapy or intolerance
* A clinical diagnosis of hypertension
* Indication for statin therapy for primary or secondary prevention of coronary artery disease
* Current or anticipated indication in ≤ 1 year for implantable cardioverter defibrillators or other metallic devices preventing cardiac magnetic resonance imaging (MRI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-04; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular mass at 12 months from baseline | 12 months

SECONDARY OUTCOMES:
a decrease in maximal ventricular wall cross sectional width | 12 months
a decrease in the incidence of nonsustained ventricular tachycardia | 12 months
a decrease in T-wave alternans | 12 months
a decrease in the volume of dense myocardial fibrosis | 12 months
parameters of diastolic function | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Sheldon, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Faculty of Medicine, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Hersi A, Giannoccaro JP, Howarth A, Exner D, Weeks S, Eitel I, Herman RC, Duff H, Ritchie D, Mcrae M, Sheldon R. Statin Induced Regression of Cardiomyopathy Trial: A Randomized, Placebo-controlled Double-blind Trial. Heart Views. 2016 Oct-Dec;17(4):129-135. doi: 10.4103/1995-705X.201784. PMID 28400935